CLINICAL TRIAL: NCT04670939
Title: the Effect of Respiratory Physiotherapy to Weaning in Invasive Mechanical Ventilation
Brief Title: Respiratory Physiotherapy in Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Canan Gursoy, Canan Gursoy, Muğla Sıtkı Koçman University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFT-CNN
Record Dates: First submitted 2019-08-18; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Respiratory Failure
Keywords: respiratory physiotherapy
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPT (Experimental)
  Interventions: Procedure: breath exercises

INTERVENTIONS:
Procedure: breath exercises — diaphragmatic breathing exercise that used during weaning is the respiratory physiotherapy

SUMMARY:
This study aimed to evaluate the effect of respiratory physiotherapy that is breathing exercise during weaning on ventilated patients in ICU.

DETAILED DESCRIPTION:
Respiratory physiotherapy is a treatment approach to increase ventilation and function in patients with acute and chronic problems and to reduce respiratory work and dyspnea.Airway cleaning techniques, lung volume-enhancing approaches, thoracic mobilization, positioning, breathing exercises and inhalation therapy are among the strategies used.

In patients with invasive MV support, respiratory physiotherapy is the position, tracheal cleaning and inhalation therapy when necessary. But breathing exercises are not indicated in the acute phase. In the process of weaning, inspiratory muscle training and breathing exercises can be used.

ELIGIBILITY:
Inclusion Criteria:

* weaning period of patients in invasive mechanical ventilation
* patients in stable hemodynamic parameters

Exclusion Criteria:

* under 18 years old
* pregnant
* non-cooperative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
weaning success | 1-7 days
  effect of respiratory physiotherapy as diaphragmatic exercise of weaning

SECONDARY OUTCOMES:
Compliance | 1-7 days
  effect of diaphragmatic exercise on compliance, diaphragmatic movement
diaphragmatic movement | 1-7 days
  effect of diaphragmatic exercise on diaphragmatic movement
arterial blood gas | 1-7 days
  effect of diaphragmatic exercise on diaphragmatic movement

CONTACTS AND LOCATIONS:
Overall Officials: Canan Gürsoy, Principal Investigator — Muğla Sıtkı Koçaman University, Training And Research Hospital
Locations (1):
- Mugla Sıtkı Kocman University Reasearch and Treaninig Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No